CLINICAL TRIAL: NCT03692026
Title: Assessment of Implant Stability in Immediate Post-extraction Implants With and Without the Application of Hyaluronic Acid and Melatonin Mixture: Randomized Clinical Trial
Brief Title: Assessment of Immediate Implant Stability When Adding Mixture of Hyaluronic Acid and Melatonin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azza Mohamed Nasr, Main investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PERIO 1405
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Immediate Dental Implant
Keywords: post-extraction implant, dental implant; melatonin; Hyaluronic acid
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: It's a Randomized Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Immediate implant placement in fresh extraction sockets with addition of Hyaluronic acid and Melatonin mixture to the implant surface, into the extraction socket and to the peri-implant area.
  Interventions: Procedure: Immediate implant placement; Drug: Hyaluronic acid and Melatonin Mixture
- Control group (Active Comparator): Immediate implant placement in fresh extraction sockets without adding any material.
  Interventions: Procedure: Immediate implant placement

INTERVENTIONS:
Procedure: Immediate implant placement — implants will be placed in freshly extraction sockets with or without application of Hyaluronic acid and Melatonin mixture.
  Other Names: early implant placement
Drug: Hyaluronic acid and Melatonin Mixture — a mixture of hyaluronic acid and melatonin will be prepared and added topically to the implant surface, extraction socket and peri-implant area for the study group
  Arms: Study group

SUMMARY:
Placing implants immediately after tooth extraction offers several advantages such as preventing bone resorption, maintaining alveolar crest width and height, reducing surgical procedures and treatment time, in addition to good esthetic results. Immediate implant placement after tooth extraction is often associated with a residual gap between the implant surface and the residual bone walls. Osseointegration between the implant surface and the surrounding osseous walls of the extraction socket should increase using materials that promote new bone formation. Since both melatonin and hyaluronic acid are thought to have a positive effect on increasing osseointegration and decreasing inflammation of the tissues; the investigators want to test if adding a mix of hyaluronic acid and melatonin to immediately implant, will give a better implant stability, decreased peri-implant bone loss and decreased post-operative pain versus immediate implant placement without adding any material.

DETAILED DESCRIPTION:
Oral rehabilitation with dental implants has become an established therapy in the past decades. Installation of implants in extraction sockets was advocated for to reduce the number of surgical procedures, time between tooth removal and installation of implant supported restoration, and to preserve the dimensions of alveolar ridge.

Scientific evidence exists demonstrating that early implantation may preserve the alveolar anatomy and that the placement of a fixture in a fresh extraction socket may help to maintain the bony crest structure. Fresh extraction sockets offer better opportunities for bone regeneration because of their particularly elevated healing potential.

Implant stability is directly related to the percentage of the bone to implant contact area (BIC). Studies had reported that osseointegration occurs following immediate implant installation in extraction sockets despite presence of marginal gap between bone and implant surface up to 4 mm. Different approaches have been introduced lately to positively enhance the healing around dental implants. One approach to enhance osseointegration of dental implants is the coating with organic components of the extracellular matrix. Recent studies have shown promising results using different organic surface modifications on dental implants, such as glycosaminoglycans, collagen and Hyaluronic acid.

Hyaluronic acid (HA) is a naturally occurring non-sulfated glycosaminoglycans which plays a role in the inflammatory process and wound healing of mineralized and non-mineralized tissues of the periodontium including granulation tissue formation and tissue remodeling. It also supports the structural and homeostatic integrity of tissues regulating properties as osmotic pressure and tissue lubrication.

It was found that coating the implants with low sulfated HA increased peri-implant bone formation around dental implants in maxillary bone compared to uncoated implants in early healing period. Another study proved that application of 1% HA associated with a collagen scaffold can improve bone formation in critical-size defects.

Furthermore, Melatonin (N-acetyl-5-methoxy tryptamine) is a substance secreted by multiple organs including the pineal gland, retina, bone marrow, the gastro-intestinal tract and the immune system. It plays an anti-inflammatory, anti-oncotic, and immunomodulatory role by scavenging free-radicals and by interacting with cell membrane and intracellular proteins. It was found to have a positive effect on new bone formation around implants as it promotes osteoblast differentiation and bone formation. Experimental evidence suggests that topical application of melatonin may be useful in oral surgery and implant dentistry, increasing BIC values and new bone formation, and so improving the success and long-term survival of the implants.

Explanation for choice of comparators:

Since both melatonin and hyaluronic acid are thought to have a positive effect on increasing osseointegration and decreasing inflammation of the tissues, the synergistic effect of both materials on the following outcomes will be investigated; implant stability, decreasing the horizontal dimensional bone loss around the implant and post-operative pain.

Aim of the study:

This study aims at assessing the effect of adding a mixture of hyaluronic acid and melatonin to the implant surface in immediate implants; regarding implant stability, peri-implant horizontal bone changes and post-operative pain, in comparison to immediate implant placement without adding any materials.

The primary objective:

Measuring the implant stability in immediate implants with hyaluronic acid and melatonin mixture, versus immediate implants placed without adding any materials.

The secondary objective:

Measuring the peri-implant horizontal bony changes and post-operative pain with topical application of hyaluronic acid and melatonin mixture to immediately placed implants, versus immediate implant placement without addition of any materials.

Trial design:

* A Randomized controlled trial.
* Unicenter study: A trial will be carried out in one hospital.
* Double blinded randomization: Neither the operator nor the patient will select the method of treatment which will be chosen by the supervisor.

Methods:

A) Participants, interventions & outcomes

. Study settings: The study will be carried out on patients attending the outpatient clinics in Oral Medicine, Diagnosis and Periodontology Department- Faculty of Oral and Dental Medicine, Cairo University-Egypt.

. Eligibility criteria:

1. Inclusion criteria 1. Age: 18-60 years old. 2. Patients with single non-restorable teeth in the inter-bicuspid area. 3. Patients with adequate bone volume for the dental implant procedure. 4. Patients who are compliant to oral hygiene measures. 5. Patients accepting to sign an informed consent to undergo the treatment.
2. Exclusion criteria:

   1. Heavy smokers.
   2. Systemic disease that contraindicates implant placement or surgical procedures.
   3. No or poor patient's compliance.
   4. Psychological problems.
   5. Periapical pathosis at the site of intervention.
   6. Pregnant females.

      * Interventions General operative procedures Eligible patients will be divided into two equal groups; study group (Immediate implant + hyaluronic acid and melatonin mixture) and control group (immediate implant alone).

   Preoperative measures (for both study and control groups): (T0)
   * All subjects will pass through phase 0 therapy (T0) (Supragingival scaling, subgingival debridement and oral hygiene instructions) before any surgical procedure is performed.
   * After 4 weeks, all subjects will be recalled for examination of their compliance to the given oral hygiene instructions; tooth brushing twice daily and chlorhexidine HCL 1.25% mouthwash (Hexitol mouthwash 100ml, ADCO, Alexandria, Egypt) twice daily.
   * Eligible patients will be randomized before being enrolled in the study.
   * The main investigator will take intraoral periapical radiographs at the time of the initial examination to confirm the diagnosis of the non-restorable tooth site using Kodak D speed films.
   * CBCT scan using OnDemand 3D (Cybermed Inc., Technoville, Gasan-dong, Geumcheon-gu, Seoul, South Korea) will be performed to record preoperative bone height and width measurements used to determine implant diameter, length and position.

   Surgical phase (T1):
   1. The main investigator will perform all procedures under local anesthesia (4% articaine with 1/200 000 adrenaline Solution) (Ubistesin forte 3M ESPE AG, ESPE Platz, D-82229 Seefeld, Germany), using a local infiltration technique for maxillary teeth or nerve block technique for mandibular teeth.
   2. A loading dose of 2 capsules of Antibiotic 875 mg of Amoxicillin and 125 mg of Clavulanic acid (2 X 1 gm Amoxicillin Clavulanate) will be given orally to the patient 1 hour before the procedure.
   3. Minimally invasive extraction of the intended tooth will be performed using Periotome (Nordent,REPC N15, US) to preserve the alveolar bone integrity, followed by irrigation of the socket with sterile saline solution and curettage to remove any remnants of the periodontal ligaments or pocket tissue.

      Intervention for study group (Group A):
   4. Melatonin and hyaluronic acid mixture will be prepared (pure melatonin will be purchased from pure bulk supplements and prepared as 5% oral gel at El-Ezaby pharmacy. Hyaluronic acid will be used in the gel form Gingigel also from El Ezaby pharmacy) The produced mixture will be added to the implant surface, into the extraction socket and in the peri-implant area.
   5. Implant will be inserted in site by flapless surgery.
   6. Primary implant stability will be measured at the day of surgery and 6 months after surgery using Ostell.
   7. Simple interrupted suture with a 5-a silk suture to approximate the labial/buccal and lingual/palatal tissues.

      Intervention for control group (Group B):

   4. Implant will be placed as in manufacturer instruction. 5. Primary implant stability will be measured at the day of surgery and 6 months after surgery using Ostell.

   6. Simple interrupted suture with a 5-a silk suture to approximate the labial/buccal and lingual/palatal tissues.

   Post-operative care: (T2) 1. Sutures will be removed after 10 days. 2. Patients in both groups will receive restoration after implant being osseointegrated.

   3. Post-operative pain will be assessed using Numerical scale for pain (NRS).

   Follow-up (T0, T1, T2):

   1. Patients will be recalled for follow up after 10 days, then every month to check on the healing of the implantation site without complications (dehiscence, inflammation, excessive pain), and to ensure that they are following proper oral hygiene measures.

   2. At the same day of surgery, implant stability will be measured using Ostell (T1).

   3. After 10 days, following suture removal, post-operative pain will be assessed using the Numerical scale of pain (NRS).

   4. After six months, implant stability will be measured again (T2) for all patients in both groups. Also, all patients will do a CBCT to compare peri-implant horizontal bony changes.

   Prosthetic phase (T3):

   1. After 6 months, implant exposure will be performed under local anaesthesia, and healing collars will be placed for 1 week before being replaced by the permanent abutment (T3).

   2. Impressions (Express, 3M ESPE, 3 M Corporate Headquarters, Maplewood, Minnesota) will be taken and fixed prosthesis will be fabricated accordingly.

   Outcomes:

   Primary outcome:
   * Implant stability:

   Implant stability quotient (ISQ) will be measured using Ostell, at the time of surgery (T1) and after 6 months (T2).

   Secondary outcomes:

   - Peri-implant horizontal bone changes: Peri-implant horizontal bone measurements in mm will be taken from pre-operative CBCT (T0) and post-osseointegration CBCT (T2) to assess the change in the horizontal bone dimensions of the peri-implant area between the two groups.

   - Post-operative pain: Post-operative pain will be recorded for all patients using the Numerical scale (NRS) of pain to compare between the values obtained for the study group and those for the control group.

ELIGIBILITY:
Inclusion Criteria:

.18-60 years old. .single non-restorable teeth in the inter-bicuspid area. .adequate bone volume for the dental implant procedure. .compliant to oral hygiene measures. .accepting to sign an informed consent to undergo the treatment.

Exclusion Criteria:

.Heavy smokers. .Systemic disease that contraindicates implant placement or surgical procedures.

* No or poor patient's compliance.
* Psychological problems.
* Periapical pathosis at the site of intervention.
* Pregnant females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Implant stability | six months
  Measuring the implant stability using Ostell device

SECONDARY OUTCOMES:
Peri-implant horizontal bone changes | six months
  peri-implant bone changes will be measured using CBCT (cone beam computed tomography)
post-operative pain | six months
  post-operative pain will be assessed using Numerical Scale of Pain (NRS). Patient describes post-operative pain on a scale from 1-10;where 1 represents the lowest value or minimum pain or no pain, while 10 represents highest value which is severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Darhous, PhD, Study Chair — Professor of Periodontology. Faculty of Oral and Dental Medicine. Cairo University; Mona Shoeib, PhD, Study Director — Professor of Periodontology. Faculty of Oral and Dental Medicine. Cairo University; Ahmed El Barbary, PhD, Study Director — Ass. Professor of Periodontology. Faculty of Oral and Dental Medicine. Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my study chair

REFERENCES:
- [Background] de Brito Bezerra B, Mendes Brazao MA, de Campos ML, Casati MZ, Sallum EA, Sallum AW. Association of hyaluronic acid with a collagen scaffold may improve bone healing in critical-size bone defects. Clin Oral Implants Res. 2012 Aug;23(8):938-42. doi: 10.1111/j.1600-0501.2011.02234.x. Epub 2011 Jun 21. PMID 21689163
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Result] Swami V, Vijayaraghavan V, Swami V. Current trends to measure implant stability. J Indian Prosthodont Soc. 2016 Apr-Jun;16(2):124-30. doi: 10.4103/0972-4052.176539. PMID 27141160
- [Result] El-Gammal MY, Salem AS, Anees MM, Tawfik MA. Clinical and Radiographic Evaluation of Immediate Loaded Dental Implants With Local Application of Melatonin: A Preliminary Randomized Controlled Clinical Trial. J Oral Implantol. 2016 Apr;42(2):119-25. doi: 10.1563/aaid-joi-D-14-00277. Epub 2015 Jun 23. PMID 26103559
- [Result] Paolantonio M, Dolci M, Scarano A, d'Archivio D, di Placido G, Tumini V, Piattelli A. Immediate implantation in fresh extraction sockets. A controlled clinical and histological study in man. J Periodontol. 2001 Nov;72(11):1560-71. doi: 10.1902/jop.2001.72.11.1560. PMID 11759868